CLINICAL TRIAL: NCT06187207
Title: Hand Acceleration Time (HAT) Assessment of the Hand's Arterial Perfusion Before and After Creating an Arteriovenous Fistula (AVF) for Dialysis: A Prospective Cohort Study
Brief Title: Hand Acceleration Time (HAT) Assessment Before and After Creating an Arteriovenous Fistula (AVF)
Acronym: HATs-ACCVAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Begoña Gonzalo Villanueva, Expert Vascular Surgeon, Hospital Universitari de Bellvitge
Other Study IDs: 2- VASC 2023
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Arteriovenous Fistula; Vascular Diseases
Keywords: Hand acceleration time; Arteriovenous Fistula; Vascular disease; Hemodialysis access-induced distal ischemia
MeSH Terms: conditions — Arteriovenous Fistula; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Candidates for AVF intervention: Patients requiring hemodialysis who are intervened for AVF creation.
  Interventions: Diagnostic Test: Hand acceleration time (HAT) measurement

INTERVENTIONS:
Diagnostic Test: Hand acceleration time (HAT) measurement — Hand Duplex Ultrasound to measure the Hand Acceleration Time (HAT)

SUMMARY:
The main objectives of this observational study are to compare the results of the sonographic parameter hand acceleration time (HAT) measured before and after creating an arteriovenous fistula (AVF) for hemodialysis and assess if it is associated with the incidence of hemodialysis access-induced distal ischemia (HAIDI).

The secondary objectives are to study the incidence of HAIDI in patients intervened for the creation of an AVF in the last 6 months, study the AVF permeability at 6 months, and study the AVF-related complications at 6 months.

DETAILED DESCRIPTION:
As the name suggests, hemodialysis access-induced distal ischemia (HAIDI) is an ischemic syndrome affecting the hand in the context of vascular access for hemodialysis. It is caused by the inability of the arterial tree to accommodate and vasodilate after the creation of an arteriovenous fistula (AVF). Furthermore, upper limbs with previously asymptomatic or paucisymptomatic arterial stenoses may suffer from higher blood flow demand after AVF is performed, thus giving rise to ischemic symptoms.

HAIDI affects 5-10% of AVF patients with a brachial fistula and less than 1% of those with a radio-cephalic fistula. The clinical presentation consists of hand hypoperfusion symptoms, which can be classified into four degrees of severity, according to Fontaine's classification. Notably, it is most commonly a chronic entity, starting approximately one month after creating the AVF.

The diagnostic work-up is often based on non-specific clinical signs and symptoms, such as coldness, paleness, trophic lesions, and absent/weak distal pulses. Complementary non-invasive tests to measure hand perfusion include determining the baseline and post-AVF compression digital pressures, digital-brachial index (DBI), plethysmography, and digital oxygen saturation. Nonetheless, no consensus exists on their reference values to diagnose HAIDI, and the definitive diagnosis often requires performing invasive procedures (arteriography).

Performing a duplex ultrasound (DUS) may be useful and provide valuable information. In the context of HAIDI, it may help us assess the proximal arterial integrity, define whether it is a high or low-flow fistula, and establish the distal arterial waveform. One interesting DUS parameter is the acceleration time (AT), which measures the time elapsed (in milliseconds) from the beginning of the arterial Doppler waveform until its systolic peak. It allows for a real-time assessment of the arterial waveform morphology.

Some authors have successfully described the reliability of the AT for lower limb assessment (pedal acceleration time, PAT), while others have used it in other arterial territories (e.g., carotid, pulmonary, and coronary arteries and the aorta). Markedly, the hand acceleration time (HAT) has also been described very recently as a potential tool to assess cardiogenic shock, subclavian iatrogenic ischemic lesions, and HAIDI. In the context of HAIDI, it may help us assess the proximal arterial integrity, define whether it is a high or low-flow fistula, and establish the distal arterial waveform. Therefore, we hypothesized that HAT is a sensitive method for detecting HAIDI in patients with an AVF.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* Both sexes
* Candidates for AVF creation for hemodialysis
* Patients who sign the informed consent form

Exclusion Criteria:

* Patients deemed unable by the investigators to understand or comply with study-related procedures
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients candidate for AVF creation for hemodialysis in the Bellvitge University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean (standard deviation, SD) HAT measured with DUS. | 24 weeks
  The HAT will be measured before the surgery for AVF creation, and at 6 and 24 weeks after the surgery in the following arteries:
  * Distal radial artery
  * Distal ulnar artery
  * Princeps pollicis artery
  * Index finger radial artery
  * First common palmar digital artery
  * Third common palmar digital artery

SECONDARY OUTCOMES:
Mean (SD) age of the participants. | Day 1
Number (percentage) of male/female participants. | Day 1
Number (percentage) of patients presenting cardiovascular risk factors of interest. | Day 1
  Cardiovascular risk factors of interest are smoking habits, arterial hypertension, diabetes mellitus, and dyslipidemia.
Number (percentage) of patients with past medical history of interest. | Day 1
  A past medical history of interest is defined as ischemic cardiopathy, heart failure, and chronic obstructive pulmonary disease.
Hemodialysis (Yes/No) at the screening visit. | Day 1
End-stage kidney disease diagnosis (Yes/No) throughout the study. | 24 weeks
Anticoagulant or antiplatelet treatment (Yes/No) throughout the study. | 24 weeks
Presence (Yes/No) of distal pulses in the upper limb. | 24 weeks
  The presence or absence of distal pulses in the upper limb will be assessed in all study visits.
Allen test (Positive/Negative) throughout the study. | Day 1
Number (percentage) of AVF types performed. | 24 weeks
  Types of AVF are:
  * Native AVF of the wrist
  * Native AVF of the elbow
  * Prosthetic AVF
Number (percentage) veins used for AVF creation. | 24 weeks
  Veins used for AVF creation can be:
  * Distal cephalic vein
  * Cephalic vein at the elbow level
  * Basilic vein at the elbow level
  * Perforating vein of the elbow
  * Axillary vein
Number (percentage) arteries used for AVF creation. | 24 weeks
  Arteries used for AVF creation can be:
  * Radial artery
  * Humeral artery
Number (percentage) of anastomosis types performed. | 24 weeks
  Types of anastomosis can be:
  * End-to-side anastomosis
  * Side-to-side anastomosis
Number (percentage) of venous outflow. | 24 weeks
  Types of venous outflow can be:
  * One anterograde vein
  * Two anterograde veins
  * One anterograde vein and 1 retrograde vein
Functional fistula (Yes/No) | 24 weeks

OTHER OUTCOMES:
Mean (SD) fistula blood flow | 6 - 24 weeks
  Other sonographic parameters besides the HAT.
Mean (SD) anastomosis length | 6 - 24 weeks
  Other sonographic parameters besides the HAT.
Mean (SD) vein diameter | 6 - 24 weeks
  Other sonographic parameters besides the HAT.
Morphology (description) of the distal radial artery spectral waveform. | 6 - 24 weeks
  Other sonographic parameters besides the HAT.

CONTACTS AND LOCATIONS:
Overall Officials: Begoña Gonzalo, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Gonzalo B, Videla S, Espinar E, Palacios S, Herranz C, Iborra Ortega E. Hand acceleration time (HAT) as a diagnostic tool in the assessment of haemodialysis access-induced distal ischaemia (HAIDI): study protocol for a prospective cohort study in the Barcelona south metropolitan area. BMJ Open. 2025 Jan 2;15(1):e093911. doi: 10.1136/bmjopen-2024-093911. PMID 39753269